CLINICAL TRIAL: NCT05604937
Title: Safety and Efficacy of Shi's Traumatology Osteopathic Manipulation for Cervicogenic Dizziness: A Randomized, Controlled, Multicenter Trial
Brief Title: Safety and Efficacy of Shi's Traumatology Osteopathic Manipulative Treatment for Cervicogenic Dizziness
Acronym: SESTOMTCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhan Yunfan (Other)
Responsible Party: Sponsor-Investigator, Zhan Yunfan, Sponsor Investigator, ShuGuang Hospital
Organization: ShuGuang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZYunfan
Record Dates: First submitted 2022-10-24; First posted 2022-11-03 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Cervicogenic Dizziness
Keywords: Cervicogenic dizziness; Vertigo; Manipulation; Osteopathic manipulative treatment
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual therapy group (Other): Patients receive Shi's traumatology osteopathic manipulative treatment twice a week and continues for 2 weeks. Receive a total of 4 manipulative treatments.
  Interventions: Other: Shi's traumatology osteopathic manipulation
- Merislon group (Other): Merislon (Betahistine Mesilate Tablets), specification 6mg, Sinopharm H20040130, Eisai (China) Pharmaceutical Co., LTD., is given to the control group, for 2 weeks, 6mg a day, three times a day.
  Interventions: Drug: Merislon

INTERVENTIONS:
Other: Shi's traumatology osteopathic manipulation — Patients receive treatment twice a week and continues for 2 weeks. Receive a total of 4 manipulative treatments. The manipulation intervention has mainly two steps: First, doctors perform soft-tissue manipulation on neck and shoulders to relax for 10 min; Second, doctors perform manipulation to reconstruct atlantoaxial joint. The strength of manipulation is based on the patient's tolerance. Do not use too much force.
  Arms: Manual therapy group
Drug: Merislon — Merislon (Betahistine Mesilate Tablets), specification 6mg, Sinopharm H20040130, Eisai (China) Pharmaceutical Co., LTD., is given to patients of the control group, for 2 weeks, 6mg a day, three times a day.
  Arms: Merislon group

SUMMARY:
This is a randomized, controlled, multi-center clinical trail to objectively evaluate safety and efficacy of shi's traumatology Osteopathic manipulative treatment for cervicogenic dizziness. Multi-center study is planned to be carried out in 4 medical institutions in Shanghai, including Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Yueyang traditional chinese and western medicine Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Baoshan traditional chinese and western medicine Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, and Shanghai General Hospital. Randomly Assigned 106 patients (18 < ages <65 ) who meet the diagnostic criteria of cervicogenic dizziness to the treatment group and the control group by a ratio of 1:1, using betahistine mesylate tablets as positive control. Observe and compare the variations of Dizziness Handicap Inventory (DHI) from baseline in two groups after 2 weeks treatment, using Dizziness Handicap Inventory (DHI) as the main efficacy index. After the end of treatment, performing 4weeks follow-up, focus to compare the recurrence rate of vertigo symptoms in the period of 4weeks follow-up after 2 weeks treatment. The safety indexes will be observed and compared, including vital sign, physical examination and adverse event, in the trail.

The electronic case Report Form (eCRF) will be used to collect and manage the study data.

The data of the primary efficacy index, DHI, patient's vertigo condition report, both use electronic patient-reported outcome (e-PRO) to collect. To ensure quality of study, this trail intends to set safeguard measures for clinical trail including setting Clinical Research Associate (CRA) to monitor study quality, evaluating efficacy by the third person, training manual therapy physicians, make access and regular and irregular assessment consistent.

DETAILED DESCRIPTION:
Recruitment Participants will be recruited from outpatients of Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Yueyang traditional chinese and western medicine Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Baoshan traditional chinese and western medicine Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, and Shanghai General Hospital. Researcher will provide both oral and written information about the trial to patients, and explain detailed information about participating in the trail, including interventions, procedures and potential adverse reactions. Written informed consent will be obtained from all participants prior to their participation. Researcher will protect the confidentiality of the participants by keeping anonymous state. Documents that have the identity participants will be kept strictly confidential. The researchers in each clinical trail center should take responsibility for medical treatment of patients and make medical decisions related to clinical trail. Ensure patients can receive effective treatment for their diseases during the clinical period or when adverse events happen.

Data management The electronic case Report Form (eCRF) will be used to collect and manage data of this trial. The primary and secondary outcomes will be collected by the eCRF.

Electronic Data Capture Data collection and Management

* CRF: CRF will be designed by data manager according to the protocol, and set up data validation rules, according to Data Validation Plan. It will be used after passing the test and being approved by sponsor.
* Data Entry: CRF data are derived from original records. Data entry personnel enter visit data of patients into Electronic Data Capture (EDC) in time, according to instructions.
* Source Data Verification (SDV): The monitor performs source data verification (SDV) to check the consistency of CRF data and source data. Issue if there has questions.
* Data Questions and Answers: Questions come from EDC logical verification system questions, auditors, data managers and other manual questions. Researchers need to timely answer questions. The data manager and the monitor will reply to the question, and may issue the question again if necessary, until the data is "clean".
* Researcher Signature: After data entering and SDV, researchers use electronic signature to review and confirm data. If data should be modified after the signature, researchers need to sign the signature again.
* Database Locking: Database locking will be signed by the main researchers, sponsor, statistical analyst and data manager. The data manager locks the database.
* Database Submitting: Database will be submitted to statistical analyst by data manager.
* CRF Archiving: Each patient's CRF will generate as a PDF electronic document for preservation
* Data Management Report: Data manager write reports of data management.
* EDC Shutdown: Data manager will shut down the database after statistical analysis completed.

External data transmission Sign external data transmission protocol and manage external data according to DMP.

Medical code Adverse events will use ICH M1: Medical Dictionary of Regulatory Activities (MedDRA) (Version 21.0 or above) to code. Drug combination use WHO ATC to classify.

Sample Size Calculation In summary of previous research reports, the effective rate of Betahistine Mesilate Tablets to vertigo patients is 60.1%. In this trail, the effective rate of the experimental group after manual therapy will be set to 85%.

Known：P1=60.1%，P2=85%，let α=0.05，β=0.20. Follow the sample size calculation formula required for completely randomized design two population rates hypothesis test to estimate. It was calculated that 47.99≈48 cases need to be observed in each group. If there are 10% to drop out, 53 patients should be included. Two groups need a total of 106 patients.

Statistical Analysis The statistical analysis will be carried out using SAS9.4 software. Except validity test uses one-side test. All of other statistical tests use a two-sided test. P < 0.05 is considered statistically significant. The primary efficacy index will be analyzed based on Intention-to-Test (ITT) and Per-Protocol set (PPS). ITT is defined as the group of patients that were randomized and had at least one treatment, and obtained the efficacy date. PPS is defined as a subset of ITT, except for incomplete drug treatment, major protocol deviation, lack of key effectiveness indexes, and other situations that are judged by blind review meeting to have a significant impact on efficacy evaluation. Main analysis model aim to analyze the variation of Vss-c score relative baseline after 2 weeks of treatment. The variation of Vss-c score relative baseline is as dependent variable, included in the baseline level for correction, and Give the overall comparison p value. Disappearing and happening time of vertigo symptom, with normal distribution, will be analyzed by independent-sample t-test. Chi-square test will be performed to analyze recurrence rate of vertigo symptom within 4 weeks of follow-up after treatment. Baseline data and descriptive statistical demographic data will calculate cases, mean, standard deviation, quartile, minimum and maximum values will be calculated for continuous variables, frequency and constituent ratio for count and grade data. Safety analysis is performed based on safety set (SS), which is defined as the group of patients who received treatment at least once and collected safety date. Adverse events will be coded according to the ICH International Medical Dictionary for Regulatory Activities (MedDRA). The frequency and incidence of adverse events/reactions, serious adverse events/reactions, and adverse events/reactions leading to shedding during treatment were calculated. Compliance analysis will be performed to calculate the percentage of compliance of patients with treatment and medication in the range of 80% to 120%. Missing date based on ITT primary efficacy indexes analysis is imputed by using LOCF method, and provide analysis results not carried forward. Other analyses are performed by using analysis results not carried forward.

ELIGIBILITY:
Inclusion Criteria:

* 18~65 years old；
* Meet diagnostic criteria of cervicogenic dizziness；
* Had cervical odontoid process deviation showed ·on CT 3D reconstruction of cervical spine or CT plain scan of atlantoaxial joint cross-section at inclusion.
* Patients had dizziness symptom at inclusion
* 31 ≤ DHI ≤ 60；
* Course of disease ≥ 1 month；
* Patients were volunteer to joint this study, and signed written informed consent.

Exclusion Criteria:

* Dizziness caused by other diseases (like otogenic, cerebral, traumatic, ophthalmogenic, neurofunctional, intracranial tumor, subclavian steal syndrome etc.)
* Cervical vertebra has fracture, dislocation, tuberculosis, acute cervical spine disc protrusion, infection, cancer;
* Patients has severe heart, liver, brain, kidney complications or other serious diseases;
* Uncontrolled hypertension grade Ⅱ or higher, or blood pressure≥160/100mmHg after antihypertensive treatment;
* Patients has a history of carotid plaque;
* Pregnancy, lactation, family planning, or patients judged not to use effective contraception.
* Patients has mental diseases;
* Has Suspected or confirmed history of alcohol or drug abuse
* Patients are afraid of Manual therapy
* Patients are allergic to betahistine mesylate tablets
* Had participated in other clinical trials within 3 months before screening
* Researchers considered Other conditions that were not appropriate to participate in the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Change of vertigo within 2 weeks of treatment | At the end of baseline (0 week), treatment for 1 week, treatment for 2 weeks and follow-up for 4 weeks.
  Change of vertigo within 2 weeks of treatment will be the primary outcome of this study. Dizziness Handicap Inventory (DHI) will be used to evaluate. The DHI consists of 25 questions, evaluated the influencing factors of vertigo or dizziness of patients from three dimensions: functional (F), emotional (E) and physical (P). Patients give scores according to their subjective conditions. Total score is DHIT (100 points), functional score is DHIF (36 points), emotional score is DHIE (36 points), and physical score is DHIP (28 points). Each question gives 4 points for answering Yes, 2 points for answering sometimes, and 0 points for answering No. The lower score means less disability. 0-30: mild vertigo; 31-60: moderate vertigo; 61-100: severe vertigo.

SECONDARY OUTCOMES:
disappearing and happening time of vertigo symptom | up to 6 weeks
  Disappearing and happening time of vertigo symptom refer to the time when vertigo happens or disappears during the whole process. It is helpful to evaluate the efficacy and recurrence rate. Disappearing time of vertigo symptom will be recorded in e-PRO system by patients.
recurrence rate of vertigo symptom within 4 weeks of follow-up after treatment | from 3rd week to 6th week
  Recurrence rate of vertigo symptom will be recorded in e-PRO system by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Wei'an Yuan, Chief, Study Chair — Shuguang Hospital Affiliated with Shanghai University of TCM
Locations (3):
- China (3):
  - Yueyang traditional Chinese and Western Medicine Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Baoshan traditional Chinese and Western Medicine Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Zhan Y, Zhang Y, Liu K, Zhao Y, Ning J, Chai Y, Kong L, Yuan W. Safety and efficacy of traditional Chinese manual therapy for cervicogenic dizziness: study protocol for a randomized, controlled, multicenter trial. Contemp Clin Trials Commun. 2024 Aug 18;41:101349. doi: 10.1016/j.conctc.2024.101349. eCollection 2024 Oct. PMID 39262903